CLINICAL TRIAL: NCT00069251
Title: Bupropion for the Treatment of Methamphetamine Dependence
Brief Title: Bupropion for the Treatment of Methamphetamine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0008-1
Record Dates: First submitted 2003-09-18; First posted 2003-09-24 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Amphetamine-Related Disorders
Keywords: amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to assess the efficacy and safety of bupropion in reducing methamphetamine use in subjects with methamphetamine dependence

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, parallel-group design study in which 100 subjects will be randomly assigned to placebo or bupropion for 12 weeks with follow-up assessments 4 weeks following treatment. Adaptive randomization will be used to balance treatment groups based on gender.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have methamphetamine dependence as determined by the DSM-IV diagnosis
* Subject must be willing to comply with study procedures.
* Ability to verbalize understanding of consent form, provide written consent, and verbalize willingness to complete study procedures
* Be able to comply with protocol requirements

Exclusion Criteria:

* Please contact site for more information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-07; Study Completion 2005-06

PRIMARY OUTCOMES:
Severity addiction
Methamphetamine use

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rawson, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - Matrix Institute on Addictions, Costa Mesa, California
  - South Bay Treatment Center, San Diego, California
  - Pacific Addiction Research Center, Honolulu, Hawaii
  - Powell Chemical Dependency Center, Des Moines, Iowa
  - University of Missouri - Kansas City, Kansas City, Missouri